CLINICAL TRIAL: NCT01669395
Title: Early Homebased Rehabilitation for Patients With Severe Heart Failure - An Intersectoral Randomized Controlled Trial
Brief Title: Severe Heart Failure and Homebased Rehabilitation - An Intersectoral Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Laura Staun Valentiner, Research and Development Physiotherapist, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-2-2012-021
Record Dates: First submitted 2012-08-14; First posted 2012-08-21 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-08

CONDITIONS: Chronic Heart Failure; Heart Failure NYHA Class II; Heart Failure NYHA Class III; Heart Failure NYHA Class IV
Keywords: Severe heart failure; Homebased rehabilitation; Physical exercise; Activities of daily living; Intersectoral Cooperation
MeSH Terms: conditions — Heart Failure; Motor Activity | interventions — Exercise; Activities of Daily Living

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early homebased rehabilitation (Experimental): After discharge from the hospital patients are offered a homebased rehabilitation program lasting 6 weeks.
  Interventions: Other: Early homebased rehabilitation after hospital admission
- control group: Ususal care (Experimental): After discharge from the hospital the patients are offered the usual symptom-oriented and preventive medical care and psychosocial support
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Early homebased rehabilitation after hospital admission — Training begins 3-5 days after discharge from hospital, performed by an occupational therapist and a physiotherapist from Gentofte Hospital in the first two weeks. From week three to six the training will be carried out by an occupational therapist and a physiotherapist from the local municipality (Gentofte municipality and Lyngby Taarbæk municipality). Training will take place at home twice a week for 6 weeks, each session lasting 45 minutes. The intervention is individualized and focuses on functional physical and compensatory training to help the patient to manage everyday life at home. A training program will be provided and the patient will be instructed to do the exercises every day
  Other Names: severe heart failure; homebased rehabilitation; physical exercise; activities of daily living
  Arms: Early homebased rehabilitation
Other: Usual care — After discharge from the hospital the patients are offered the usual symptom-oriented and preventive medical care and psychosocial support
  Arms: control group: Ususal care

SUMMARY:
The purpose of this study is to investigate the effect of an early, coordinated rehabilitation intervention for patients with severe heart failure in NYHA class III and IV with a ejection fraction of <40% of normal cardiac function measured on frequency of readmissions, physical ability and participation in activities of daily living and quality of life.

DETAILED DESCRIPTION:
Approximately 400,000 Danes live today with heart disease. Disease severity is crucial for patients quality of life. Patients with severe heart disease often struggle with everyday life, characterized by reduced physical capacity, tendency to depression and anxiety to perform everyday activities that may provoke symptoms.

A large proportion of patients who are offered cardiac rehabilitation deselect that offer. Of the patients who do participate, more than 50% stop the rehabilitation ahead of time. A large group of patients with severe heart failure and classified in NYHA Class III and IV, deselect the offer because of lack of energy to participate in cardiac rehabilitation or is when specified by a medical assessment discharged from the hospital without the offer of training or any other form of rehabilitation.

The offer of rehabilitation for patients with severe heart failure is lacking as it is today. This study assesses the effectiveness of an early home based rehabilitation program that complements the general psycho-social support, symptom-oriented and preventive medical treatment that these patients always have the option to get.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the Gentofte Hospital due to heart failure.
* Patients with a functional equivalent to NYHA grade III or IV
* Patients with ejection fraction <40%
* Patients who score between10-15 in the total score for question 3 dealing with physical functioning in SF-36 questionnaire on health status
* Patients who lives in Gentofte Municipality or Lyngby Tårbæk Municipality.
* Patients who can speak and understand Danish

Exclusion Criteria:

* Patients with cognitive and psychological problems that prevents cooperation (aphasia, dementia, severe depression).
* Patients with terminal illness with expected death within a year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-09 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Readmission due to heart failure | assessed one year after inclusion

SECONDARY OUTCOMES:
Physical capacity | Assessed at baseline, after 6 weeks, after 6 month and after one year
  measured by the Morton Mobility Index, Timed Up & Go and Modified Sit to Stand Test
Activity of Daily Living | Assessed at baseline, after 6 weeks, after 6 month and after one year
  Recorded at an ADL interview to assess the performance of everyday activities
Number of total hospital admissions | at baseline, after 6 weeks, after 6 month and after one year
Exercise Compliance | at baseline, after 6 weeks, after 6 month and after one year
  registration of exercise
Anxiety and depression | at baseline, after 6 weeks, after 6 month and after one year
  measured by Hospital Anxiety and Depression Scale (HAD)
Quality of life | at baseline, after 6 weeks, after 6 month and after one year
  measured by The Minnesota Living with Heart Failure Questionnaire
Number of patients who starts outpatient cardiac rehabilitation after intervention (municipality or hospital) | at 6 weeks, after 6 month and after one year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Occupational Therapy and Physiotherapy, Copenhagen University Hospital Gentofte,, Copenhagen, Gentofte, Denmark